CLINICAL TRIAL: NCT02044211
Title: Blended Collaborative Care for Heart Failure and Co-Morbid Depression
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Bruce Rollman, Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HL114016 (NIH)
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Heart Failure, Systolic; Depression; Cardiovascular Disease
Keywords: Heart Failure, Systolic; Depressive Disorder; Depressive Disorder, Major; Mood Disorder
MeSH Terms: conditions — Heart Failure, Systolic; Depression; Cardiovascular Diseases; Depressive Disorder; Depressive Disorder, Major; Mood Disorders

STUDY DESIGN:
Intervention Model Description: "Blended" intervention: Blended, centralized, nurse-provided, telephone-delivered collaborative care for both heart failure and depression;
  Collaborative care for heart failure: Blended, centralized, nurse-provided, telephone-delivered collaborative care for heart failure alone
  Usual Care: PCPs usual care for heart failure and depression; and
  Non-Depressed comparison cohort (randomly sampled, not randomized).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Collaborative Care for Heart Failure + Depression (Active Comparator): Collaborative care program for heart failure and depression involving a nurse care manager providing counseling and treatment advice via telephone
  Interventions:
  Behavioral:
  Counseling for heart failure self-care Counseling for depression
  Drug:
  Pharmacotherapy for heart failure Pharmacotherapy for depression
  Interventions: Behavioral: Collaborative Care for Heart Failure; Behavioral: Collaborative Care for Depression
- Collaborative Care for Heart Failure Only (Active Comparator): Collaborative care program for heart failure and depression involving a nurse care manager providing counseling and treatment advice via telephone
  Interventions:
  Behavioral:
  Counseling for heart failure self-care Usual care for depression
  Drug:
  Pharmacotherapy for heart failure
  Usual Care for depression
  Interventions: Behavioral: Collaborative Care for Heart Failure
- Usual Care for Heart Failure and Depression (No Intervention): Control group will receive their doctors' usual care for heart failure and depression
- Non-Depressed Comparison Cohort (No Intervention): Control group will receive their doctors' usual care for heart failure

INTERVENTIONS:
Behavioral: Collaborative Care for Heart Failure — Nurse care managers will provide patients with education for their heart failure to facilitate self-management for their condition. In addition, the nurse will telephone the patient to review with their medical history, medications, diet, activity and sleep patterns, and plans for follow-up medical appointments, and offer basic care coordination relative to heart failure care including assistance attaining authorization for home health services in concert with the patient's primary care physician (PCP), and follow-up appointments.
  After case review with a study internist, the care manager may send treatment recommendations to the patient's physician(s) regarding guideline-indicated care. Afterwards, the care manager will telephone the patient approximately every other week to monitor and promote adherence with recommended care, and suggest adjustments in treatment as applicable following discussion with the clinical team and notification of the patient's PCP and cardiologist.
  Arms: Collaborative Care for Heart Failure + Depression; Collaborative Care for Heart Failure Only
Behavioral: Collaborative Care for Depression — The care manager will telephone patients randomized to "blended" care patient to review their psychiatric history including use of antidepressant pharmacotherapy, herbal supplements, and alcohol possibly used to self-medicate depressive symptoms; provide basic psychoeducation about depression and its impact on cardiac disease; recommend various self-management strategies (e.g., sufficient rest and exercise); and describe treatment options. They will include: (1) use of a workbook or computer program to enhance patients' understanding and ability to self-care; (2) initiation or adjustment of antidepressant pharmacotherapy prescribed under their primary care physicians' direction; or (3) referral to a local mental health specialist. The nurse will then telephone the patient to monitor symptoms and pharmacotherapy use, practice skills imparted through workbook assignments, promote adherence with recommended care, and suggest adjustments in treatment as applicable.
  Arms: Collaborative Care for Heart Failure + Depression

SUMMARY:
Depression is highly prevalent among patients with heart failure (HF) and associated with lower levels of health-related quality of life and physical functioning, and higher risk of rehospitalization and mortality, and higher health costs. This Project will compare the effectiveness of a "blended" telephone-delivered collaborative care intervention for treating both HF and depression to: (1) collaborative care for HF-alone ("enhanced usual care"; eUC); and (2) doctors' "usual care" for depression (UC). If proven effective and cost-effective, the potentially more powerful, scalable, efficient "blended" care approach for treating HF and co-morbid depression could have profound implications for improving chronic illness care and stimulate development of "blended" interventions for treating other clusters of related medical conditions.

DETAILED DESCRIPTION:
Heart failure (HF) is an important public health problem that affects approximately 6.6 million Americans. Despite improvements in cardiac care, it remains the leading cause for hospitalization among Medicare patients and the only major cardiovascular disease whose mortality rate has remained essentially unchanged over the past decade. This failure to improve HF outcomes may be due, in part, to unrecognized and/or inadequately treated depression that is highly prevalent in HF patients. Yet while new HF treatment guidelines advocate routine screening for depression, this recommendation is unlikely to be widely adopted without trial evidence that depression care improves outcomes and efficient methods to provide it.

"Collaborative care" strategies are being increasingly utilized to improve care for HF and other chronic medical conditions, and we recently demonstrated its clinical and cost-effectiveness at treating depression following coronary artery bypass graft surgery. Yet it may be impractical for health care delivery systems to support separate treatment programs for HF and depression. Thus we are encouraged by emerging evidence indicating "blended" collaborative care strategies that target both psychiatric and physical conditions produce greater improvements in mood symptoms and control of cardiovascular risk factors than programs focused solely on depression to propose testing a novel adaptation that could be provided in routine care.

The Specific Aims of this Project are to: (1) evaluate the effectiveness of a telephone-delivered "blended" collaborative care intervention for treating HF and depression that could be adopted into routine clinical practice if proven effective; and (2) advance our understanding of the moderators and mediators of depression treatment on clinical outcomes. We will screen hospitalized patients with systolic HF for depression, and then randomize 625 who screen positive and have at least a moderately elevated level of depressive symptoms at two-weeks following hospital discharge to either: (1) collaborative care for treating both HF and depression ("blended"); (2) collaborative care for treating HF alone (enhanced usual care (eUC)); or (3) their doctors' "usual care" (UC). Additionally, we will enroll 125 non-depressed HF patients to better evaluate the benefits derived from treating depression (total N=750). Our co-primary hypotheses will test whether "blended" collaborative care can produce at 12-months follow-up a: (A) 0.50 effect size (ES) or greater improvement in health-related quality of life (HRQoL) vs. UC; and (B) 0.30 ES or greater improvement in HRQoL vs. eUC. Secondary hypotheses will evaluate the effects of our "blended" intervention on mood, functional status, adherence with guideline-consistent care, incidence of cardiovascular events, health care utilization, and costs.

Improving chronic illness care for medically complex patients is one of the major challenges facing medicine today. We propose to test the effectiveness of an innovative, efficient, scalable, and sustainable intervention that could transform the way HF and other cardiovascular disorders are treated in routine practice.

ELIGIBILITY:
Inclusion Criteria:

1. Systolic heart failure (documented ejection fraction ≤ 40%).
2. HF symptoms meeting criteria for New York Heart Association (NYHA) classes II, III or IV.
3. Inpatient two-item Patient Health Questionnaire (PHQ-2) screen-positive for depression; or PHQ-2 screen negative for depression and PHQ-9 <5 if non-depressed control.
4. PHQ-9 ≥ 10 when reassessed two-weeks following hospital discharge, or PHQ-9 <5 if non-depressed control.
5. No cognitive impairment (as documented in the record, use of donepezil or similar medications for treating cognitive impairment, or the Montreal Cognitive Assessment).
6. Able to be evaluated and treated for depression as an outpatient.
7. English speaking, not illiterate, or possessing any other communication barrier.
8. Have a household telephone.

Exclusion Criteria:

1. Receiving active treatment for a mood or anxiety disorder from a mental health specialist.
2. Unstable medical condition as indicated by history, physical, and/or laboratory findings.
3. Presence of non-cardiovascular conditions likely to be fatal within 12 months (e.g., cancer).
4. Organic mood syndromes, including those secondary to medical illness or drugs.
5. Active suicidal ideation.
6. Current or history of psychotic illness.
7. Current or history of bipolar illness according to patient self-report, past medical history, and diagnostic criteria.
8. Current alcohol or other substance abuse as evidenced by chart review and the AUDIT-C questionnaire.
9. Age ≤ 21 years.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 756 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Medical Outcomes Study (MOS) 12-Item Short Form Health Survey Mental Component Summary (SF-12 MCS) | 12-Months Follow-Up
  Mental Health-Related Quality of Life

SECONDARY OUTCOMES:
Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | 12-Month Follow-Up
  Disease-Specific Health-Related Quality of Life
Hamilton Rating Scale for Depression (17-Item) | 12-Months Follow-Up
  Mood symptoms
Incidence of Rehospitalization | 12-Month Follow-Up
Mortality | 12-Month Follow-Up
  All-Cause and Cardiovascular Mortality
Health Care Costs | 12-Month Follow-Up
  Claims data
Employment | 12-Months Follow-Up

CONTACTS AND LOCATIONS:
Overall Officials: Bruce L. Rollman, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Deveney TK, Belnap BH, Mazumdar S, Rollman BL. The prognostic impact and optimal timing of the Patient Health Questionnaire depression screen on 4-year mortality among hospitalized patients with systolic heart failure. Gen Hosp Psychiatry. 2016 Sep-Oct;42:9-14. doi: 10.1016/j.genhosppsych.2016.06.005. Epub 2016 Jun 30. PMID 27638965
- [Background] Schuster JM, Belnap BH, Roth LH, Rollman BL. The Checklist Manifesto in action: integrating depression treatment into routine cardiac care. Gen Hosp Psychiatry. 2016 May-Jun;40:1-3. doi: 10.1016/j.genhosppsych.2016.01.005. Epub 2016 Jan 22. No abstract available. PMID 26916974
- [Background] Herbeck Belnap B, Anderson A, Abebe KZ, Ramani R, Muldoon MF, Karp JF, Rollman BL. Blended Collaborative Care to Treat Heart Failure and Comorbid Depression: Rationale and Study Design of the Hopeful Heart Trial. Psychosom Med. 2019 Jul/Aug;81(6):495-505. doi: 10.1097/PSY.0000000000000706. PMID 31083056
- [Background] Rollman BL. Exercise and Cognitive Training to Improve Neurocognitive Outcomes in Patients With Heart Failure: Can Cardiac Rehabilitation Deliver? Am J Geriatr Psychiatry. 2019 Aug;27(8):820-822. doi: 10.1016/j.jagp.2019.05.001. Epub 2019 May 6. No abstract available. PMID 31151835
- [Derived] Bober T, Guhl EN, Rothenberger S, Jeong K, Abebe KZ, Holber J, Anderson AM, Magnani JW, Johnson AE, Rollman BL. Impact of Neighborhood Factors on Heart Failure Outcomes: Secondary Analysis From the Hopeful Heart Trial. JACC Adv. 2025 Oct;4(10 Pt 2):102146. doi: 10.1016/j.jacadv.2025.102146. Epub 2025 Sep 14. PMID 40953541
- [Derived] Carrillo A, Belnap BH, Rothenberger SD, Feldman R, Rollman BL, Celano CM. Psychosocial predictors of health behavior adherence in heart-failure patients with comorbid depression: a secondary analysis of the Hopeful Heart trial. BMC Psychol. 2024 Jun 4;12(1):328. doi: 10.1186/s40359-024-01816-4. PMID 38835104
- [Derived] Sadlonova M, Chavanon ML, Kwonho J, Abebe KZ, Celano CM, Huffman J, Herbeck Belnap B, Rollman BL. Depression Subtypes in Systolic Heart Failure: A Secondary Analysis From a Randomized Controlled Trial. J Acad Consult Liaison Psychiatry. 2023 Sep-Oct;64(5):444-456. doi: 10.1016/j.jaclp.2023.03.008. Epub 2023 Mar 29. PMID 37001642
- [Derived] Holber JP, Abebe KZ, Huang Y, Jakicic JM, Anderson AM, Belnap BH, Rollman BL. The Relationship Between Objectively Measured Step Count, Clinical Characteristics, and Quality of Life Among Depressed Patients Recently Hospitalized With Systolic Heart Failure. Psychosom Med. 2022 Feb-Mar 01;84(2):231-236. doi: 10.1097/PSY.0000000000001034. PMID 34724453
- [Derived] Rollman BL, Anderson AM, Rothenberger SD, Abebe KZ, Ramani R, Muldoon MF, Jakicic JM, Herbeck Belnap B, Karp JF. Efficacy of Blended Collaborative Care for Patients With Heart Failure and Comorbid Depression: A Randomized Clinical Trial. JAMA Intern Med. 2021 Oct 1;181(10):1369-1380. doi: 10.1001/jamainternmed.2021.4978. PMID 34459842
- See also: Center for Research on Health Care — https://www.gim-crhc.pitt.edu/
- See also: Related trial of collaborative care for treating depression following coronary artery bypass graft (CABG) surgery — http://hopefulheart.pitt.edu/
- See also: Center for Behavioral Health and Smart Technology — http://www.healthtech.pitt.edu/index.php